CLINICAL TRIAL: NCT04067492
Title: An Open-label, Single-dose, Active-controlled Randomized Phase IIa Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RPH-104 (RPH-104/L04018) Administered at Different Doses to Patients With Acute Gout Attack
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Evaluation of RPH-104 Administered at Different Doses to Patients With Acute Gout Attack
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: In view of the continuing insufficient patient recruitment in the study due to the difficult epidemiological situation and the need for rational allocation of company resources, as well as based on the results of the interim analysis.
Sponsor: R-Pharm (Industry)
Collaborators: Covance (Industry); Unimed Laboratories (Industry); Data Matrix Solutions (Other); Center of Pharmaceutical Analytics LLC (Industry); OCT LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL04018054
Record Dates: First submitted 2019-08-05; First posted 2019-08-26 (Actual); Results first posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-03

CONDITIONS: Gout Attack
Keywords: hyperuricemia; acute arthritis; gouty arthritis; gout
MeSH Terms: conditions — Hyperuricemia; Arthritis, Gouty; Gout | interventions — Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- RPH - 4 mg (Experimental): Subjects randomized to receive RPH-104, 4 mg, subcutaneous single-dose injection. In order to administer RPH-104 at the dose of 4 mg, 0.1 mL of RPH-104 solution is injected.
  Interventions: Drug: RPH - 104
- RPH - 20 mg (Experimental): Subjects randomized to receive RPH-104, 20 mg, subcutaneous single-dose injection. In order to administer RPH-104 at the dose of 20 mg, 0.5 mL of RPH-104 solution is injected.
  Interventions: Drug: RPH - 104
- RPH - 40 mg (Experimental): Subjects randomized to receive RPH-104, 40 mg, subcutaneous single-dose injection. In order to administer RPH-104 at the dose of 40 mg, 1 mL of RPH-104 solution is injected.
  Interventions: Drug: RPH - 104
- RPH - 80 mg (Experimental): Subjects randomized to receive RPH-104, 80 mg, subcutaneous single-dose injection. In order to administer RPH-104 at the dose of 80 mg, 2 mL (whole vial) of RPH-104 solution is injected.
  Interventions: Drug: RPH - 104
- RPH - 160 mg (Experimental): Subjects randomized to receive RPH-104, 160 mg, two subcutaneous injections of 80 mg administered at different injection sites. (1 vial of 2mL solution per each site)
  Interventions: Drug: RPH - 104
- Voltaren® (diclofenac) (Active Comparator): Subjects randomized to receive Voltaren® (diclofenac) orally with water at the dose 50 mg thrice daily for 3 days (150 mg total daily dose), then 25 mg thrice daily for 9 days (75 mg total daily dose)
  Interventions: Drug: Voltaren®

INTERVENTIONS:
Drug: RPH - 104 — solution for subcutaneous administration 40 mg/mL, 2 mL in the 4-mL glass vial
  Arms: RPH - 160 mg; RPH - 20 mg; RPH - 4 mg; RPH - 40 mg; RPH - 80 mg
Drug: Voltaren® — Enteric-coated tablets, 25 mg and 50 mg
  Other Names: Diclofenac
  Arms: Voltaren® (diclofenac)

SUMMARY:
The primary goal of the study was to evaluate the parameters of efficacy, pharmacokinetics, pharmacodynamics, safety and tolerability of a single dose of RPH-104 in adult patients with acute gout attack.

DETAILED DESCRIPTION:
The study consisted of two periods:

Period 1. In Study Period 1, eligible patients were enrolled in a group of 22 patients and randomized to receive either RPH-104 4 mg or Voltaren® (diclofenac) in the 15:7 ratio (15 RPH-104: 7 Voltaren® (diclofenac)). In order to prevent damage to the gastric and duodenal mucosa caused by Voltaren® (diclofenac), all patients receiving Voltaren® (diclofenac) had to simultaneously take Ortanol® (omeprazole) 20 mg, orally (1 capsule) daily before breakfast throughout the course of Voltaren® (diclofenac) treatment

Period 2. Upon completion of the enrollment of 22 patients, Study Period 2 started. In Period 2, newly enrolled patients were randomly assigned to one of 5 treatment groups: RPH-104 20 mg, 40 mg, 80 mg and 160 mg and active control (Voltaren® (diclofenac)). It was planned to include 14 patients in the RPH-104 groups in Period 2, and 7 patients in the Voltaren® (diclofenac) group.

The enrollment of patients in Period 1 and Period 2 was sequential. There was no pause between the enrollment of patients in Period 1 and Period 2. The study design included screening (24 hours), 11 visits to the study site, and a phone call at the end of the 60-day follow-up period.

Total number of patients which were planned to be enrolled for the study: 85 (15 patients in the group of treatment with RPH-104 4 mg and 14 patients in the each of the other treatment groups). Due to the low patient recruitment rate in the study and the negative impact of the COVID-19 pandemic on the recruitment, at the decision of the sponsor, an interim analysis of the data of 47 patients included in the study as of November 2020 was carried out in order to assess the feasibility of continuing recruitment and further conducting the study.

Patients who did not tolerate pain were allowed to receive a rescue medication, triamcinolone acetonide 40 mg intramuscularly, to intensify therapy 2 hours after the test product was administered. If the attack recurred after the use of the rescue medication, treatment was carried out in accordance with the standard practice of the hospital.

The primary efficacy endpoints were evaluated 72 hours after the end of administration of the test drug. The secondary efficacy endpoints were evaluated for 45 days of the treatment period and follow-up. The safety parameters were evaluated for 60 days of the treatment period and follow-up. Total duration of the study for a volunteer was not more than 70 days.

ELIGIBILITY:
Inclusion Criteria:

* 1. The subject has given his / her informed consent to participate in this study; the Informed Consent Form has been signed both by the patient and the Investigator;
* 2. Established diagnosis of gout according to Gout Classification Criteria established by the American College of Rheumatology (ACR) and European League against Rheumatism (EULAR) in 2015;
* 3. Pain in at least one joint at the screening and immediately prior to initiation of therapy with the study drugs, with intensity 50 mm to 100 mm according to the Visual Analogue Scale (VAS);
* 4. Development of acute gout attack within 120 hours (5 days) prior to the randomization date;
* 5. History of 1 or more acute gout attacks prior to the Screening Visit;
* 6.The patients receiving uric acid-lowering drugs should continue receiving these drugs at a constant dose for at least 4 weeks prior to enrolment to the study and throughout the entire study period; the patients not receiving uric acid-lowering drugs may start receiving this treatment after the end of the study;
* 7. Body mass index ≤40 kg/m2;
* 8. QTcF interval ≤450 msec for male subjects and ≤470 msec for females on ECG at the screening;
* 9. For women of child-bearing potential: negative result of the serum pregnancy test performed at the screening;
* 10. The consent of a woman of child-bearing potential, as well as of a man who has female partners of child-bearing potential, to abstain from sexual intercourses or to use effective birth control methods throughout the entire study period and for 60 days after RPH-104 administration (if the patient received RPH-104);
* 11. The patient is able to fulfil the requirements of the Study Protocol as judged by the Investigator

Exclusion Criteria:

* 1. The patient received therapy with ibuprofen in a dose of up to 400 mg inclusive within 4 hours or >400 mg within 8 hours prior to randomization.
* 2. The patient received therapy with diclofenac in a dose of up to 50 mg inclusive within 8 hours or >50 mg within 24 hours prior to randomization.
* 3. The patient received any other non-steroidal anti-inflammatory drug (NSAID) within 24 hours prior to the randomization;
* 4.The patient received opioids within 48 hours prior to the randomization;
* 5. The patient received metamizole or metamizole-containing drugs within 12 hours prior to the randomization;
* 6. The patient received any drug with analgesic activity (including paracetamol) within 6 hours prior to the randomization;
* 7. The patient received a long-acting NSAID (half-life ≥24 hours) within 5 half-life periods or 1 month prior to the randomization whichever is longer;
* 8. The patient received extended-release naproxen, meloxicam, nabumetone, celecoxib, etoricoxib or indomethacin within 5 days prior to the randomization;
* 9 . The patient received corticosteroids (including their intra-articular administration and inhalations) within 4 weeks prior to the randomization;
* 10. The patient received colchicine within 7 days prior to the randomization;
* 11. Intolerance or contraindications for NSAID use;
* 12. Contraindications for the use of Ortanol® capsules 20 mg;
* 13. Chronic heart failure functional class II-IV (classification of NYHA);
* 14. A history of or current clinically significant ventricular arrhythmias or clinically significant atrial tachyarrhythmias;
* 15. Unstable angina or stable exercise-induced angina of functional class III or IV;
* 16. Secondary gout, chemotherapy-induced gout, lead- or transplantation-induced gout;
* 17. Rheumatoid arthritis, confirmed or suspected infectious septic arthritis or any other type of acute inflammatory arthritis;
* 18. Clinically significant renal impairment determined based on creatinine clearance (estimated using the Cockcroft-Gault equation) <60 mL/min, or patients on hemodialysis;
* 19. Blood coagulation disorders; history of gastrointestinal bleedings or perforation;
* 20. Pregnant or breast-feeding women;
* 21. Elective surgery or major surgical intervention (minor surgical procedures, such as catheter placement or bone marrow biopsy, are not exclusion criteria) within 14 days before the first dose of the investigational medicinal product;
* 22. Current or suspected HIV-infection, HBsAg, Hepatitis C Virus antibodies (HCVAb), other acute or chronic bacterial, fungal or viral infections at the moment of subject's enrolment to the study;
* 23. Presence of any risk factors for tuberculosis based on the results of assessment using Tuberculosis Risk Assessment Questionnaire at the screening or confirmed tuberculosis or any other infectious disease of the lungs or bronchi based on findings of the chest X-ray exam in two views performed within 3 months prior to the screening visit, or the need for using therapy with tuberculosis medications, such as isoniazid in the course of the study;
* 24. Neutropenia, leukopenia, or thrombocytopenia determined based on the following laboratory parameters assessed during the screening:

  1. Absolute neutrophil count (ANC) <1.5 x 10^9/L;
  2. White blood cell count <4.0 х 10^9/L
  3. Platelet count <150 х 10^9/L;
* 25. Immunization with live vaccines within 3 months prior to the subject's enrolment to the study or planned vaccination within 60 days after the expected date of the first dose of the test drug;
* 26. History of allergic reactions to biologicals, Voltaren® (diclofenac) or Ortanol® (omeprazole);
* 27. Contraindications for subcutaneous, intramuscular, intravenous or intra-articular injections;
* 28. History of malignancy (except for patients with localized in situ basal cell carcinoma of the skin or in situ cervical cancer, who can be enrolled to the study immediately after the therapy for this disease), unless it is in remission for ≥5 years, as well as patients who are being examined for cancer or patients with suspected malignancy;
* 29. A condition or disease, which, in the Investigator's opinion, could put the patient's safety at risk or affect the test drug safety assessment;
* 30. Any other conditions and diseases, such as uncontrolled diabetes mellitus, uncontrolled hypertension, congestive heart failure, exacerbation of peptic ulcer disease, clinically significant liver diseases, kidney diseases, uncontrolled thyroid dysfunction, unhealed wounds, ulcers or bone fractures, psychiatric disorders, uncontrolled epilepsy, drug dependence, which could prevent the patient from complying with this Study Protocol.
* 31. The patient received biologicals or investigational medicinal products within 5 half-life periods of these drugs or 3 month prior to the randomization whichever is longer;
* 32. Blood donation or blood loss of ≥400 mL within 8 weeks prior to the randomization.
* 33. The patient was already randomized in this clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — R-Pharm
Locations (11):
- Russia (11):
  - Moscow City State Healthcare Institution "O.M. Filatov Municipal Clinical Hospital No. 15" of the Moscow Department of Healthcare, Moscow
  - State Budgetary Healthcare Institution of Moscow City "Municipal Clinical Hospital No.1 named after N.I. Pirogov" of Moscow Department of Healthcare, Moscow
  - Federal State Autonomous Educational Institution of Higher Education "I.M. Sechenov First Moscow State Medical University of the Ministry of Health of the Russian Federation (Sechenov University), Moscow
  - State Budgetary Healthcare Institution of Moscow City "Municipal Clinical Hospital No.52" of Moscow Department of Healthcare, Moscow
  - State Budgetary Institution of Healthcare of Nizhny Novgorod region "City Clinical hospital #13 of Avozavodskiy district", Nizhny Novgorod
  - Federal State Budgetary Education Institution of Higher Education "Orenburg State Medical University" under Ministry of Healthcare of Russian Federation, Orenburg
  - St. Petersburg State Budgetary Healthcare Institution "Clinical Rheumatological Hospital No.25", Saint Petersburg
  - State Budget Institution "Saint Petersburg Research Insitute of emergency care named after I.I. Dzhanelidze, Saint Petersburg
  - Limited Liability company "Scientific Research Center Eco-safety", Saint Petersburg
  - State Insitution of healthcare "Tula regional clinical dermatovenerologic dispensary", Tula
  - State Autonomous Healthcare Institution of the Yaroslavl Region "N.V. Solovyev Clinical Emergency Hospital", Yaroslavl

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was conducted at 11 clinical sites in Russian Federation. 54 subjects were screened and 47 subjects were enrolled (randomized) and treated, 44 subjects completed the study.
  The Safety Population and Efficacy Population included data from all 47 randomized patients to assess safety, treatment efficacy and pharmacodynamics.
Groups:
- RPH - 4 mg: RPH-104, 4 mg, subcutaneous single-dose injection. 0.1 mL of 40 mg/mL RPH-104 solution is injected.
- RPH - 20 mg: RPH-104, 20 mg, subcutaneous single-dose injection. 0.5 mL of 40 mg/mL RPH-104 solution is injected.
- RPH - 40 mg: RPH-104, 40 mg, subcutaneous single-dose injection.
  1 mL of 40 mg/mL RPH-104 solution is injected.
- RPH - 80 mg: RPH-104, 80 mg, subcutaneous single-dose injection. 2 mL (whole vial) of 40 mg/mL RPH-104 solution is injected.
- RPH - 160 mg: RPH-104, 160 mg, two subcutaneous injections of 80 mg administered at different injection sites.
  1 vial of 2mL 40 mg/mL solution per each site
- Voltaren® (Diclofenac): Voltaren® (diclofenac) orally with water at the dose 50 mg thrice daily for 3 days (150 mg total daily dose), then 25 mg thrice daily for 9 days (75 mg total daily dose) (Voltaren®: Enteric-coated tablets, 25 mg and 50 mg)
Period: Overall Study
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac)
Started | 15 | 6 | 6 | 6 | 5 | 9
Completed | 15 | 5 | 6 | 5 | 5 | 8
Not Completed | 0 | 1 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Not completed — closure of city borders because of COVID-19 quarantine | 0 | 1 | 0 | 0 | 0 | 0
Not completed — COVID-19 epidemiological situation | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac) | Total
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 5 | 9 | 47
Age, Continuous [Mean (Full Range); unit: years] | 52.3 [31 to 63] | 51.7 [46 to 60] | 42.8 [34 to 57] | 56.5 [41 to 78] | 53.6 [50 to 59] | 52.2 [42 to 61] | 51.5 [31 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 0 | 0 | 2 | 3
  Male | 15 | 5 | 6 | 6 | 5 | 7 | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian/White | 15 | 6 | 6 | 6 | 5 | 9 | 47
  Race: other | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disease duration [Mean (Full Range); unit: years] | 8.13 [0.9 to 17.2] | 7.65 [0.1 to 17.3] | 8.04 [2.4 to 19.4] | 9.16 [0.9 to 15.9] | 13.55 [7.4 to 29.3] | 6.41 [0.1 to 12.5] | 8.82 [0.1 to 29.3]
Exact number of affected joints [Mean (Full Range); unit: number (of joints)] | 5.3 [1 to 23] | 3.0 [1 to 5] | 5.7 [1 to 25] | 2.7 [1 to 5] | 6.2 [2 to 16] | 3.0 [1 to 7] | 4.32 [1 to 25]

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity in the Assessed Joint 72 Hours After the Initiation of Treatment in Comparison to Baseline
Description: Change in pain intensity in the assessed joint 72 hours after the initiation of treatment with the test drug measured using the Visual Analogue Scale (VAS) in comparison to baseline. VAS is a hard copy 100 mm scale with the indications: "Absence of pain" on the left side of the scale (0 mm point) and "The most severe pain ever experienced" on the right side of the scale (100 mm point)) The better outcome would be "Absence of pain", the worse outcome would be "The most severe pain ever experienced".
Time Frame: Baseline and Day 4 (72 hours after the initiation of treatment with the test drug)
Population: The baseline observation carried forward method (BOCF) was used to impute missing data for the main efficacy analysis. Missing patient data were replaced with baseline values from the time of patient discontinuation or use of the rescue medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm (VAS scale)
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 5 | 9
mm (VAS scale) | -7.88 [-22.26 to 6.50] | -38.56 [-60.39 to -16.72] | -19.80 [-41.83 to 2.22] | -33.39 [-55.53 to -11.24] | -30.55 [-54.46 to -6.64] | -36.51 [-55.11 to -17.90]
Statistical Analysis 1: Comparison: RPH - 4 mg vs Voltaren® (Diclofenac); It was assumed that the sample size would allow constructing a 95% CI around the mean change in pain intensity at 72 hours after the start of the investigational product use in each group with an accuracy of 30 mm change in pain intensity and would reveal statistically significant differences between the groups in pairwise comparisons, without control for type I error for multiple comparisons, taking into account the type I error α = 5%, if the difference between the compared groups is ≥ 20 mm; Test type: Other — The study was planned to randomize 85 patients: 15 patients in the RPH-104 4 mg group, and 14 patients in the RPH-104 20 mg, 40 mg, 80 mg and 160 mg groups each, a total of 14 patients in the Voltaren® (diclofenac) group. The sample size was calculated assuming a standard deviation of 26 mm for change in pain intensity at 72 hours; p = 0.1331, ANCOVA — p-value, group; Mean Difference (Final Values) = 28.63, 95% CI 2-sided [4.21 to 53.05] — Adjusted mean difference. Comparison with the control group [RPH-104 - Diclofenac]
Statistical Analysis 2: Comparison: RPH - 20 mg vs Voltaren® (Diclofenac); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.1331, ANCOVA — p-value, group; Mean Difference (Final Values) = -2.05, 95% CI 2-sided [-30.60 to 26.50] — Adjusted mean difference. Comparison with the control group [RPH-104 - Diclofenac]
Statistical Analysis 3: Comparison: RPH - 40 mg vs Voltaren® (Diclofenac); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.1331, ANCOVA — p-value, group; Mean Difference (Final Values) = 16.70, 95% CI 2-sided [-12.67 to 46.08] — Adjusted mean difference. Comparison with the control group [RPH-104 - Diclofenac]
Statistical Analysis 4: Comparison: RPH - 80 mg vs Voltaren® (Diclofenac); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.1331, ANCOVA — p-value, group; Mean Difference (Final Values) = 3.12, 95% CI 2-sided [-25.10 to 31.33] — Adjusted mean difference. Comparison with the control group [RPH-104 - Diclofenac]
Statistical Analysis 5: Comparison: RPH - 160 mg vs Voltaren® (Diclofenac); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.1331, ANCOVA — p-value, group; Mean Difference (Final Values) = 5.96, 95% CI 2-sided [-24.22 to 36.14] — Adjusted mean difference. Comparison with the control group [RPH-104 - Diclofenac]

2. Secondary Outcome: Change in Pain Intensity in the Assessed Joint in 15, 30, 45 Minutes, 1, 1.5, 2, 4, 8, 24, 48, 72 Hours, on Days 5, 6, 10, 15, 18, 22, 29 and 45 Following the Initiation of Treatment and Compared to Baseline
Description: Change in pain intensity in the assessed joint in 15, 30, 45 minutes, 1, 1.5, 2, 4, 8, 24, 48, 72 hours, on Days 5, 6, 10, 15, 18, 22, 29 and 45 following the initiation of treatment with the test drug measured using the Visual Analogue Scale (VAS) and compared to baseline. VAS is a hard copy 100 mm scale with the indications: "Absence of pain" on the left side of the scale (0 mm point) and "The most severe pain ever experienced" on the right side of the scale (100 mm point)) The better outcome would be "Absence of pain", the worse outcome would be "The most severe pain ever experienced".
Time Frame: Baseline and 15, 30, 45 minutes, 1, 1.5, 2, 4, 8, 24, 48, 72 hours, on Days 5, 6, 10, 15, 18, 22, 29 and 45 after the initiation of treatment
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mm (VAS scale)
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 5 | 9
mm (VAS scale)
  Day 1/15 minutes | -2.00 [-6.38 to 2.38] | -6.97 [-13.81 to -0.14] | -5.91 [-12.76 to 0.94] | -1.52 [-8.39 to 5.34] | -5.75 [-13.23 to 1.74] | -3.78 [-9.44 to 1.88]
  Day 1/30 minutes | -10.00 [-16.81 to -3.19] | -14.16 [-24.87 to -3.45] | -6.43 [-17.15 to 4.29] | -5.19 [-15.92 to 5.54] | -10.57 [-22.30 to 1.16] | -5.45 [-14.24 to 3.35]
  Day 1/45 minutes | -16.20 [-24.71 to -7.69] | -16.14 [-29.55 to -2.73] | -7.91 [-21.33 to 5.51] | -9.36 [-22.78 to 4.07] | -11.77 [-26.45 to 2.92] | -8.56 [-19.55 to 2.43]
  Day 1/ 1 hour | -19.67 [-30.12 to -9.21] | -15.81 [-32.30 to 0.69] | -11.76 [-28.27 to 4.74] | -12.52 [-29.03 to 3.99] | -15.99 [-34.06 to 2.09] | -12.67 [-26.17 to 0.83]
  Day 1/ 1.5 hours | -22.47 [-32.96 to -11.97] | -15.14 [-31.70 to 1.42] | -21.26 [-37.82 to -4.70] | -14.69 [-31.26 to 1.88] | -17.79 [-35.92 to 0.35] | -13.67 [-27.22 to -0.12]
  Day 1/ 2 hours | -22.07 [-33.65 to -10.48] | -25.14 [-43.42 to -6.86] | -24.63 [-42.92 to -6.34] | -13.86 [-32.15 to 4.44] | -19.59 [-39.62 to 0.44] | -20.56 [-35.52 to -5.60]
  Day 1/ 4 hours | -21.87 [-34.63 to -9.10] | -27.27 [-47.43 to -7.12] | -21.44 [-41.61 to -1.28] | -14.36 [-34.52 to 5.81] | -20.35 [-42.43 to 1.73] | -22.67 [-39.15 to -6.19]
  Day 1/ 8 hours | -14.20 [-27.05 to -1.35] | -29.61 [-49.89 to -9.32] | -18.93 [-39.22 to 1.36] | -16.52 [-36.82 to 3.77] | -25.35 [-47.57 to -3.13] | -25.67 [-42.26 to -9.08]
  Day 2 | -10.60 [-23.27 to 2.07] | -37.77 [-57.77 to -17.78] | -20.94 [-40.95 to -0.94] | -25.52 [-45.53 to -5.52] | -30.35 [-52.25 to -8.44] | -30.34 [-46.69 to -13.98]
  Day 3 | -3.33 [-16.21 to 9.54] | -35.77 [-56.10 to -15.45] | -27.94 [-48.28 to -7.61] | -34.69 [-55.03 to -14.35] | -30.15 [-52.41 to -7.88] | -38.67 [-55.29 to -22.05]
  Day 4 | -6.67 [-20.38 to 7.05] | -38.77 [-60.43 to -17.11] | -18.91 [-40.58 to 2.76] | -34.52 [-56.19 to -12.85] | -30.75 [-54.47 to -7.02] | -38.12 [-55.83 to -20.40]
  Day 5 | -4.73 [-18.62 to 9.15] | -31.27 [-53.20 to -9.35] | -13.64 [-35.57 to 8.28] | -35.86 [-57.79 to -13.92] | -31.35 [-55.36 to -7.33] | -42.78 [-60.71 to -24.86]
  Day 6 | -4.80 [-18.42 to 8.82] | -34.44 [-55.95 to -12.93] | -12.43 [-33.95 to 9.09] | -22.86 [-44.38 to -1.33] | -29.15 [-52.71 to -5.58] | -42.45 [-60.04 to -24.86]
  Day 10 | -6.73 [-21.29 to 7.82] | -37.27 [-60.26 to -14.29] | -12.43 [-35.42 to 10.57] | -23.52 [-46.52 to -0.53] | -29.15 [-54.33 to -3.96] | -37.78 [-56.57 to -18.99]
  Day 15 | -4.13 [-18.21 to 9.94] | -41.77 [-64.00 to -19.55] | -12.41 [-34.64 to 9.82] | -12.69 [-34.93 to 9.55] | -28.95 [-53.30 to -4.60] | -38.34 [-56.51 to -20.16]
  Day 18 | -4.07 [-18.18 to 10.05] | -42.61 [-64.90 to -20.31] | -12.74 [-35.04 to 9.55] | -12.69 [-34.99 to 9.61] | -29.75 [-54.17 to -5.33] | -28.45 [-46.67 to -10.22]
  Day 22 | -3.20 [-17.43 to 11.03] | -44.61 [-67.08 to -22.14] | -13.58 [-36.05 to 8.90] | -12.69 [-35.17 to 9.79] | -28.35 [-52.96 to -3.73] | -30.34 [-48.71 to -11.97]
  Day 29 | -4.07 [-18.36 to 10.23] | -44.94 [-67.52 to -22.36] | -13.58 [-36.16 to 9.01] | -12.69 [-35.28 to 9.90] | -17.95 [-42.68 to 6.79] | -23.89 [-42.35 to -5.43]
  Day 45 | -2.60 [-16.67 to 11.48] | -46.94 [-69.17 to -24.71] | -13.58 [-35.81 to 8.66] | -12.69 [-34.93 to 9.55] | -19.75 [-44.09 to 4.60] | -23.34 [-41.51 to -5.16]

3. Secondary Outcome: Proportion of Patients Who Assessed the Response to Therapy With the Test Drug as "Excellent" or "Good"
Description: Proportion of patients who assessed the response to therapy with the test drug as "Excellent" or "Good" in 15, 30, 45 minutes, 1, 1.5, 2, 4, 8, 24, 48, 72 hours, on Days 5, 6, 10, 15, 18, 22, 29 and 45 following the initiation of treatment with the test drug.
  The patient's response to therapy was assessed in the form of frequency tables by assessment point and therapy group. The rates of the response were specified in the evaluation form as: "Excellent", "Good", "Fair", "Weak", "Poor" (where "excellent" represents the best possible response to treatment and "poor" indicates the worst treatment response).
Time Frame: 15, 30, 45 minutes, 1, 1.5, 2, 4, 8, 24, 48, 72 hours, on Days 5, 6, 10, 15, 18, 22, 29 and 45 after the initiation of treatment with the test drug
Population: The table shows the frequencies and proportions (%) of the number of valid observations. Values after the use of rescue medication and after withdrawal were imputed as failure.
Measure: Count of Participants; unit: Participants
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 5 | 9
Participants
  Day 1/15 minutes: number analyzed (Participants) | 15 | 4 | 6 | 6 | 5 | 9
  Day 1/15 minutes | 0 | 1 | 0 | 1 | 0 | 1
  Day 1/30 minutes: number analyzed (Participants) | 15 | 4 | 6 | 6 | 5 | 9
  Day 1/30 minutes | 2 | 1 | 0 | 1 | 0 | 2
  Day 1/45 minutes: number analyzed (Participants) | 15 | 4 | 6 | 6 | 5 | 9
  Day 1/45 minutes | 3 | 1 | 0 | 2 | 0 | 2
  Day 1/ 1 hour: number analyzed (Participants) | 15 | 4 | 6 | 6 | 5 | 9
  Day 1/ 1 hour | 3 | 0 | 0 | 2 | 0 | 1
  Day 1/ 1.5 hours: number analyzed (Participants) | 15 | 4 | 6 | 6 | 5 | 9
  Day 1/ 1.5 hours | 3 | 0 | 1 | 1 | 0 | 1
  Day 1/ 2 hours: number analyzed (Participants) | 15 | 4 | 6 | 6 | 5 | 9
  Day 1/ 2 hours | 3 | 0 | 1 | 1 | 0 | 1
  Day 1/ 4 hours: number analyzed (Participants) | 15 | 4 | 6 | 6 | 5 | 9
  Day 1/ 4 hours | 2 | 0 | 2 | 1 | 1 | 2
  Day 1/ 8 hours: number analyzed (Participants) | 15 | 4 | 6 | 6 | 5 | 9
  Day 1/ 8 hours | 2 | 1 | 2 | 1 | 2 | 4
  Day 2: number analyzed (Participants) | 15 | 4 | 6 | 6 | 5 | 9
  Day 2 | 1 | 0 | 2 | 1 | 2 | 2
  Day 3: number analyzed (Participants) | 15 | 4 | 6 | 6 | 5 | 9
  Day 3 | 1 | 1 | 2 | 1 | 2 | 5
  Day 4: number analyzed (Participants) | 15 | 4 | 6 | 6 | 5 | 9
  Day 4 | 1 | 1 | 1 | 3 | 2 | 6
  Day 5: number analyzed (Participants) | 15 | 4 | 6 | 6 | 5 | 9
  Day 5 | 1 | 1 | 1 | 3 | 2 | 6
  Day 6: number analyzed (Participants) | 15 | 4 | 6 | 6 | 5 | 9
  Day 6 | 1 | 2 | 1 | 2 | 2 | 6
  Day 10: number analyzed (Participants) | 15 | 3 | 6 | 6 | 5 | 9
  Day 10 | 1 | 1 | 1 | 2 | 2 | 6
  Day 15: number analyzed (Participants) | 15 | 4 | 6 | 6 | 5 | 9
  Day 15 | 1 | 2 | 1 | 1 | 2 | 6
  Day 18: number analyzed (Participants) | 15 | 3 | 6 | 6 | 5 | 9
  Day 18 | 1 | 1 | 1 | 1 | 2 | 4
  Day 22: number analyzed (Participants) | 15 | 4 | 6 | 6 | 5 | 9
  Day 22 | 0 | 2 | 1 | 1 | 2 | 5
  Day 29: number analyzed (Participants) | 15 | 4 | 6 | 6 | 5 | 9
  Day 29 | 1 | 2 | 1 | 1 | 1 | 3
  Day 45: number analyzed (Participants) | 15 | 3 | 6 | 6 | 5 | 9
  Day 45 | 0 | 1 | 1 | 1 | 1 | 3

4. Secondary Outcome: Change in the Rate of Swelling of the Assessed Joint Evaluated After the Initiation of Treatment With the Test Drug
Description: Change in the rate of swelling of the assessed joint evaluated in 24, 48, 72 hours, on Days 5, 6, 10, 15, 18, 22, 29 and 45 following the initiation of treatment with the test drug compared to baseline. The rates of swelling were specified in the evaluation form as: "absence" = no swelling, "mild" = palpable swelling, "moderate" = visible swelling, "severe" = bulging outside the joint (where "severe" represented the worst possible degree of swelling and "absence" was the best outcome).
Time Frame: Baseline and 24, 48, 72 hours, on Days 5, 6, 10, 15, 18, 22, 29 and 45 following the initiation of treatment with the test drug
Population: It should be noted that estimates following the use of the rescue medication or a prohibited analgesic were not included in the descriptive statistics, therefore, the number of patients with analyzable data in treatment groups decreased over time.
Measure: Count of Participants; unit: Participants
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 5 | 9
Participants
  Baseline: absence | 0 | 0 | 0 | 0 | 0 | 0
  Baseline: mild | 1 | 0 | 0 | 0 | 0 | 1
  Baseline: moderate | 9 | 3 | 2 | 4 | 1 | 5
  Baseline: severe | 5 | 3 | 4 | 2 | 4 | 3
  Day 2/ 24 hours: number analyzed (Participants) | 12 | 5 | 6 | 5 | 4 | 8
  Day 2/ 24 hours: absence | 1 | 0 | 0 | 1 | 1 | 0
  Day 2/ 24 hours: mild | 2 | 2 | 1 | 1 | 1 | 5
  Day 2/ 24 hours: moderate | 8 | 3 | 2 | 3 | 2 | 3
  Day 2/ 24 hours: severe | 1 | 0 | 3 | 0 | 0 | 0
  Day 3/ 48 hours: number analyzed (Participants) | 2 | 5 | 5 | 4 | 3 | 7
  Day 3/ 48 hours: absence | 1 | 1 | 0 | 3 | 1 | 2
  Day 3/ 48 hours: mild | 1 | 3 | 1 | 0 | 0 | 5
  Day 3/ 48 hours: moderate | 0 | 1 | 1 | 1 | 2 | 0
  Day 3/ 48 hours: severe | 0 | 0 | 3 | 0 | 0 | 0
  Day 4/ 72 hours: number analyzed (Participants) | 2 | 5 | 3 | 3 | 3 | 7
  Day 4/ 72 hours: absence | 1 | 2 | 1 | 3 | 1 | 4
  Day 4/ 72 hours: mild | 1 | 2 | 0 | 0 | 1 | 2
  Day 4/ 72 hours: moderate | 0 | 1 | 0 | 0 | 1 | 1
  Day 4/ 72 hours: severe | 0 | 0 | 2 | 0 | 0 | 0
  Day 5: number analyzed (Participants) | 2 | 4 | 2 | 3 | 3 | 7
  Day 5: absence | 1 | 2 | 1 | 3 | 1 | 4
  Day 5: mild | 1 | 1 | 0 | 0 | 1 | 2
  Day 5: moderate | 0 | 1 | 0 | 0 | 1 | 1
  Day 5: severe | 0 | 0 | 1 | 0 | 0 | 0
  Day 6: number analyzed (Participants) | 2 | 4 | 2 | 2 | 3 | 7
  Day 6: absence | 1 | 2 | 1 | 2 | 1 | 4
  Day 6: mild | 1 | 2 | 0 | 0 | 2 | 3
  Day 6: moderate | 0 | 0 | 1 | 0 | 0 | 0
  Day 6: severe | 0 | 0 | 0 | 0 | 0 | 0
  Day 10: number analyzed (Participants) | 2 | 3 | 2 | 2 | 3 | 4
  Day 10: absence | 1 | 3 | 1 | 2 | 2 | 4
  Day 10: mild | 1 | 0 | 0 | 0 | 1 | 0
  Day 10: moderate | 0 | 0 | 1 | 0 | 0 | 0
  Day 10: severe | 0 | 0 | 0 | 0 | 0 | 0
  Day 15: number analyzed (Participants) | 1 | 4 | 1 | 1 | 3 | 6
  Day 15: absence | 1 | 4 | 1 | 1 | 2 | 6
  Day 15: mild | 0 | 0 | 0 | 0 | 1 | 0
  Day 15: moderate | 0 | 0 | 0 | 0 | 0 | 0
  Day 15: severe | 0 | 0 | 0 | 0 | 0 | 0
  Day 18: number analyzed (Participants) | 1 | 3 | 1 | 1 | 3 | 2
  Day 18: absence | 1 | 2 | 1 | 1 | 2 | 2
  Day 18: mild | 0 | 1 | 0 | 0 | 1 | 0
  Day 18: moderate | 0 | 0 | 0 | 0 | 0 | 0
  Day 18: severe | 0 | 0 | 0 | 0 | 0 | 0
  22: number analyzed (Participants) | 1 | 4 | 1 | 1 | 2 | 2
  22: absence | 1 | 3 | 1 | 1 | 1 | 2
  22: mild | 0 | 1 | 0 | 0 | 1 | 0
  22: moderate | 0 | 0 | 0 | 0 | 0 | 0
  22: severe | 0 | 0 | 0 | 0 | 0 | 0
  29: number analyzed (Participants) | 1 | 4 | 1 | 1 | 1 | 4
  29: absence | 1 | 4 | 1 | 1 | 0 | 4
  29: mild | 0 | 0 | 0 | 0 | 1 | 0
  29: moderate | 0 | 0 | 0 | 0 | 0 | 0
  29: severe | 0 | 0 | 0 | 0 | 0 | 0
  45: number analyzed (Participants) | 1 | 3 | 1 | 1 | 1 | 4
  45: absence | 0 | 3 | 1 | 1 | 0 | 4
  45: mild | 1 | 0 | 0 | 0 | 1 | 0
  45: moderate | 0 | 0 | 0 | 0 | 0 | 0
  45: severe | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Change in the Rate of Tenderness of the Assessed Joint Evaluated After the Initiation of Treatment With the Test Drug
Description: Change in the rate of tenderness of the assessed joint evaluated in 24, 48, 72 hours, on Days 5, 6, 10, 15, 18, 22, 29 and 45 following the initiation of treatment with the test drug compared to baseline. Tenderness degrees: "absent" = no tenderness, "mild" = tenderness when touched, "moderate" = pain and flinching, "severe" = pain, flinching and withdrawal of the limb (where "severe" represents the worst possible degree of tenderness and "absent" is the best outcome).
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 5 | 9
Participants
  Baseline: absence | 0 | 0 | 0 | 0 | 0 | 0
  Baseline: mild | 1 | 1 | 0 | 0 | 0 | 0
  Baseline: moderate | 12 | 4 | 3 | 4 | 2 | 6
  Baseline: severe | 2 | 1 | 3 | 2 | 3 | 3
  Day 2/ 24 hours: number analyzed (Participants) | 12 | 5 | 6 | 5 | 4 | 8
  Day 2/ 24 hours: absence | 1 | 0 | 0 | 1 | 2 | 0
  Day 2/ 24 hours: mild | 4 | 5 | 3 | 1 | 1 | 6
  Day 2/ 24 hours: moderate | 6 | 0 | 1 | 3 | 1 | 2
  Day 2/ 24 hours: severe | 1 | 0 | 2 | 0 | 0 | 0
  Day 3/ 48 hours: number analyzed (Participants) | 2 | 5 | 5 | 4 | 3 | 7
  Day 3/ 48 hours: absence | 1 | 0 | 0 | 1 | 1 | 1
  Day 3/ 48 hours: mild | 1 | 5 | 2 | 2 | 2 | 6
  Day 3/ 48 hours: moderate | 0 | 0 | 1 | 1 | 0 | 0
  Day 3/ 48 hours: severe | 0 | 0 | 2 | 0 | 0 | 0
  Day 4/ 72 hours: number analyzed (Participants) | 2 | 5 | 3 | 3 | 3 | 7
  Day 4/ 72 hours: absence | 1 | 2 | 0 | 2 | 1 | 3
  Day 4/ 72 hours: mild | 1 | 3 | 1 | 1 | 2 | 4
  Day 4/ 72 hours: moderate | 0 | 0 | 1 | 0 | 0 | 0
  Day 4/ 72 hours: severe | 0 | 0 | 1 | 0 | 0 | 0
  Day 5: number analyzed (Participants) | 2 | 4 | 2 | 3 | 3 | 7
  Day 5: absence | 1 | 2 | 1 | 3 | 1 | 3
  Day 5: mild | 1 | 2 | 0 | 0 | 1 | 4
  Day 5: moderate | 0 | 0 | 0 | 0 | 1 | 0
  Day 5: severe | 0 | 0 | 1 | 0 | 0 | 0
  Day 6: number analyzed (Participants) | 2 | 4 | 2 | 2 | 3 | 7
  Day 6: absence | 1 | 2 | 1 | 2 | 1 | 4
  Day 6: mild | 1 | 2 | 0 | 0 | 2 | 3
  Day 6: moderate | 0 | 0 | 1 | 0 | 0 | 0
  Day 6: severe | 0 | 0 | 0 | 0 | 0 | 0
  Day 10: number analyzed (Participants) | 2 | 3 | 2 | 2 | 3 | 4
  Day 10: absence | 1 | 3 | 1 | 2 | 2 | 4
  Day 10: mild | 1 | 0 | 0 | 0 | 1 | 0
  Day 10: moderate | 0 | 0 | 1 | 0 | 0 | 0
  Day 10: severe | 0 | 0 | 0 | 0 | 0 | 0
  Day 15: number analyzed (Participants) | 1 | 4 | 1 | 1 | 3 | 6
  Day 15: absence | 1 | 3 | 1 | 1 | 2 | 5
  Day 15: mild | 0 | 1 | 0 | 0 | 1 | 1
  Day 15: moderate | 0 | 0 | 0 | 0 | 0 | 0
  Day 15: severe | 0 | 0 | 0 | 0 | 0 | 0
  Day 18: number analyzed (Participants) | 1 | 3 | 1 | 1 | 3 | 2
  Day 18: absence | 1 | 3 | 1 | 1 | 2 | 1
  Day 18: mild | 0 | 0 | 0 | 0 | 1 | 1
  Day 18: moderate | 0 | 0 | 0 | 0 | 0 | 0
  Day 18: severe | 0 | 0 | 0 | 0 | 0 | 0
  22: number analyzed (Participants) | 1 | 4 | 1 | 1 | 2 | 2
  22: absence | 0 | 3 | 1 | 1 | 1 | 1
  22: mild | 1 | 1 | 0 | 0 | 1 | 1
  22: moderate | 0 | 0 | 0 | 0 | 0 | 0
  22: severe | 0 | 0 | 0 | 0 | 0 | 0
  29: number analyzed (Participants) | 1 | 4 | 1 | 1 | 1 | 4
  29: absence | 1 | 3 | 1 | 1 | 1 | 3
  29: mild | 0 | 1 | 0 | 0 | 0 | 1
  29: moderate | 0 | 0 | 0 | 0 | 0 | 0
  29: severe | 0 | 0 | 0 | 0 | 0 | 0
  45: number analyzed (Participants) | 1 | 3 | 1 | 1 | 1 | 4
  45: absence | 0 | 3 | 1 | 1 | 0 | 4
  45: mild | 1 | 0 | 0 | 0 | 1 | 0
  45: moderate | 0 | 0 | 0 | 0 | 0 | 0
  45: severe | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Change in the Rate of Erythema of the Assessed Joint Evaluated After the Initiation of Treatment With the Test Drug
Description: Change in the rate of erythema of the assessed joint evaluated in 24, 48, 72 hours, on Days 5, 6, 10, 15, 18, 22, 29 and 45 following the initiation of treatment with the test drug compared to baseline.The rates of "erythema" were specified as "absence", "presence", "impossible to evaluate".
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 5 | 9
Participants
  Baseline: absence | 3 | 0 | 0 | 0 | 0 | 2
  Baseline: presence | 12 | 6 | 6 | 5 | 5 | 7
  Baseline: evaluation impossible | 0 | 0 | 0 | 1 | 0 | 0
  Day 2/ 24 hours: number analyzed (Participants) | 12 | 5 | 6 | 5 | 4 | 8
  Day 2/ 24 hours: absence | 5 | 2 | 1 | 1 | 2 | 2
  Day 2/ 24 hours: presence | 7 | 3 | 4 | 4 | 2 | 6
  Day 2/ 24 hours: evaluation impossible | 0 | 0 | 1 | 0 | 0 | 0
  Day 3/ 48 hours: number analyzed (Participants) | 2 | 5 | 5 | 4 | 3 | 7
  Day 3/ 48 hours: absence | 2 | 4 | 2 | 3 | 1 | 5
  Day 3/ 48 hours: presence | 0 | 1 | 2 | 1 | 2 | 2
  Day 3/ 48 hours: evaluation impossible | 0 | 0 | 1 | 0 | 0 | 0
  Day 4/ 72 hours: number analyzed (Participants) | 2 | 5 | 3 | 3 | 3 | 7
  Day 4/ 72 hours: absence | 2 | 4 | 1 | 3 | 2 | 7
  Day 4/ 72 hours: presence | 0 | 1 | 2 | 0 | 1 | 0
  Day 4/ 72 hours: evaluation impossible | 0 | 0 | 0 | 0 | 0 | 0
  Day 5: number analyzed (Participants) | 2 | 4 | 2 | 3 | 3 | 7
  Day 5: absence | 2 | 4 | 1 | 3 | 3 | 7
  Day 5: presence | 0 | 0 | 1 | 0 | 0 | 0
  Day 5: evaluation impossible | 0 | 0 | 0 | 0 | 0 | 0
  Day 6: number analyzed (Participants) | 2 | 4 | 2 | 2 | 3 | 7
  Day 6: absence | 2 | 4 | 1 | 2 | 3 | 7
  Day 6: presence | 0 | 0 | 1 | 0 | 0 | 0
  Day 6: evaluation impossible | 0 | 0 | 0 | 0 | 0 | 0
  Day 10: number analyzed (Participants) | 2 | 3 | 2 | 2 | 3 | 4
  Day 10: absence | 2 | 3 | 1 | 2 | 3 | 4
  Day 10: presence | 0 | 0 | 1 | 0 | 0 | 0
  Day 10: evaluation impossible | 0 | 0 | 0 | 0 | 0 | 0
  Day 15: number analyzed (Participants) | 1 | 4 | 1 | 1 | 3 | 6
  Day 15: absence | 1 | 4 | 1 | 1 | 3 | 6
  Day 15: presence | 0 | 0 | 0 | 0 | 0 | 0
  Day 15: evaluation impossible | 0 | 0 | 0 | 0 | 0 | 0
  Day 18: number analyzed (Participants) | 1 | 3 | 1 | 1 | 3 | 2
  Day 18: absence | 1 | 3 | 1 | 1 | 3 | 2
  Day 18: presence | 0 | 0 | 0 | 0 | 0 | 0
  Day 18: evaluation impossible | 0 | 0 | 0 | 0 | 0 | 0
  22: number analyzed (Participants) | 1 | 4 | 1 | 1 | 2 | 2
  22: absence | 1 | 4 | 1 | 1 | 2 | 2
  22: presence | 0 | 0 | 0 | 0 | 0 | 0
  22: evaluation impossible | 0 | 0 | 0 | 0 | 0 | 0
  29: number analyzed (Participants) | 1 | 4 | 1 | 1 | 1 | 4
  29: absence | 1 | 3 | 1 | 1 | 1 | 4
  29: presence | 0 | 1 | 0 | 0 | 0 | 0
  29: evaluation impossible | 0 | 0 | 0 | 0 | 0 | 0
  45: number analyzed (Participants) | 1 | 3 | 1 | 1 | 1 | 4
  45: absence | 1 | 3 | 1 | 1 | 1 | 4
  45: presence | 0 | 0 | 0 | 0 | 0 | 0
  45: evaluation impossible | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Change in the Rate of Movement Restrictions in the Specified Timeframes After Initiation of Treatment
Description: Change in the rate of movement restrictions in the assessed joint evaluated in 24, 48, 72 hours, on Days 5, 6, 10, 15, 18, 22, 29 and 45 following the initiation of treatment with the test drug compared to baseline. For the assessment, the categorical scale consistent with the Form for evaluation (Investigator's Assessment) of the restriction of movements was used. The rates of movement restrictions (amplitude of movements) were specified in the evaluation form as "1 - Normal range", "2 - Slightly limited range", " 3 - Moderately limited range" ,"4 - Severely limited range" and "5 - Joint movement is impossible " (where higher score means worse outcome).
Time Frame: Baseline and in 24, 48, 72 hours, on Days 5, 6, 10, 15, 18, 22, 29 and 45 following the initiation of treatment with the test drug
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 5 | 9
Participants
  Baseline: 1 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline: 2 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline: 3 | 5 | 2 | 1 | 3 | 2 | 6
  Baseline: 4 | 9 | 4 | 5 | 2 | 2 | 3
  Baseline: 5 | 1 | 0 | 0 | 1 | 1 | 0
  Day 2/ 24 hours: number analyzed (Participants) | 12 | 5 | 6 | 5 | 4 | 8
  Day 2/ 24 hours: 1 | 1 | 0 | 0 | 0 | 0 | 0
  Day 2/ 24 hours: 2 | 0 | 1 | 0 | 2 | 2 | 4
  Day 2/ 24 hours: 3 | 7 | 3 | 3 | 2 | 1 | 3
  Day 2/ 24 hours: 4 | 3 | 1 | 2 | 1 | 1 | 1
  Day 2/ 24 hours: 5 | 1 | 0 | 1 | 0 | 0 | 0
  Day 3/ 48 hours: number analyzed (Participants) | 2 | 5 | 5 | 4 | 3 | 7
  Day 3/ 48 hours: 1 | 0 | 0 | 0 | 1 | 1 | 1
  Day 3/ 48 hours: 2 | 1 | 5 | 2 | 2 | 1 | 4
  Day 3/ 48 hours: 3 | 1 | 0 | 1 | 1 | 0 | 2
  Day 3/ 48 hours: 4 | 0 | 0 | 1 | 0 | 1 | 0
  Day 3/ 48 hours: 5 | 0 | 0 | 1 | 0 | 0 | 0
  Day 4/ 72 hours: number analyzed (Participants) | 2 | 5 | 3 | 3 | 3 | 7
  Day 4/ 72 hours: 1 | 1 | 2 | 1 | 2 | 1 | 2
  Day 4/ 72 hours: 2 | 0 | 3 | 0 | 1 | 1 | 5
  Day 4/ 72 hours: 3 | 1 | 0 | 1 | 0 | 0 | 0
  Day 4/ 72 hours: 4 | 0 | 0 | 1 | 0 | 1 | 0
  Day 4/ 72 hours: 5 | 0 | 0 | 0 | 0 | 0 | 0
  Day 5: number analyzed (Participants) | 2 | 4 | 2 | 3 | 3 | 7
  Day 5: 1 | 1 | 3 | 1 | 3 | 1 | 3
  Day 5: 2 | 0 | 1 | 0 | 0 | 1 | 4
  Day 5: 3 | 1 | 0 | 0 | 0 | 0 | 0
  Day 5: 4 | 0 | 0 | 1 | 0 | 1 | 0
  Day 5: 5 | 0 | 0 | 0 | 0 | 0 | 0
  Day 6: number analyzed (Participants) | 2 | 4 | 2 | 2 | 3 | 7
  Day 6: 1 | 1 | 3 | 1 | 2 | 1 | 5
  Day 6: 2 | 0 | 1 | 0 | 0 | 1 | 2
  Day 6: 3 | 1 | 0 | 0 | 0 | 0 | 0
  Day 6: 4 | 0 | 0 | 1 | 0 | 1 | 0
  Day 6: 5 | 0 | 0 | 0 | 0 | 0 | 0
  Day 10: number analyzed (Participants) | 2 | 3 | 2 | 2 | 3 | 4
  Day 10: 1 | 1 | 3 | 1 | 2 | 2 | 3
  Day 10: 2 | 0 | 0 | 0 | 0 | 0 | 1
  Day 10: 3 | 1 | 0 | 0 | 0 | 0 | 0
  Day 10: 4 | 0 | 0 | 1 | 0 | 1 | 0
  Day 10: 5 | 0 | 0 | 0 | 0 | 0 | 0
  Day 15: number analyzed (Participants) | 1 | 4 | 1 | 1 | 3 | 6
  Day 15: 1 | 1 | 3 | 1 | 1 | 2 | 5
  Day 15: 2 | 0 | 1 | 0 | 0 | 0 | 1
  Day 15: 3 | 0 | 0 | 0 | 0 | 1 | 0
  Day 15: 4 | 0 | 0 | 0 | 0 | 0 | 0
  Day 15: 5 | 0 | 0 | 0 | 0 | 0 | 0
  Day 18: number analyzed (Participants) | 1 | 3 | 1 | 1 | 3 | 2
  Day 18: 1 | 0 | 3 | 1 | 1 | 2 | 2
  Day 18: 2 | 1 | 0 | 0 | 0 | 0 | 0
  Day 18: 3 | 0 | 0 | 0 | 0 | 1 | 0
  Day 18: 4 | 0 | 0 | 0 | 0 | 0 | 0
  Day 18: 5 | 0 | 0 | 0 | 0 | 0 | 0
  Day 22: number analyzed (Participants) | 1 | 4 | 1 | 1 | 2 | 2
  Day 22: 1 | 0 | 3 | 1 | 1 | 1 | 2
  Day 22: 2 | 1 | 1 | 0 | 0 | 0 | 0
  Day 22: 3 | 0 | 0 | 0 | 0 | 1 | 0
  Day 22: 4 | 0 | 0 | 0 | 0 | 0 | 0
  Day 22: 5 | 0 | 0 | 0 | 0 | 0 | 0
  Day 29: number analyzed (Participants) | 1 | 4 | 1 | 1 | 1 | 4
  Day 29: 1 | 0 | 3 | 1 | 1 | 0 | 4
  Day 29: 2 | 1 | 0 | 0 | 0 | 0 | 0
  Day 29: 3 | 0 | 1 | 0 | 0 | 1 | 0
  Day 29: 4 | 0 | 0 | 0 | 0 | 0 | 0
  Day 29: 5 | 0 | 0 | 0 | 0 | 0 | 0
  Day 45: number analyzed (Participants) | 1 | 3 | 1 | 1 | 1 | 4
  Day 45: 1 | 0 | 3 | 1 | 1 | 0 | 4
  Day 45: 2 | 0 | 0 | 0 | 0 | 0 | 0
  Day 45: 3 | 1 | 0 | 0 | 0 | 1 | 0
  Day 45: 4 | 0 | 0 | 0 | 0 | 0 | 0
  Day 45: 5 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Time to Achieve the 50% Decrease in Pain Intensity in the Assessed Joint Relative to the Baseline
Description: Time to achieve the 50% decrease in pain intensity in the assessed joint relative to the baseline VAS level.
  VAS is a hard copy 100 mm scale with the indications: "Absence of pain" on the left side of the scale (0 mm point) and "The most severe pain ever experienced" on the right side of the scale (100 mm point)). The better outcome would be "Absence of pain", the worse outcome would be "The most severe pain ever experienced".
Time Frame: Baseline and one of the pain intensity measurements in accordance with the schedule: 15, 30, 45 minutes, 1, 1.5, 2, 4, 8, 24, 48, 72 hours, on Days 5, 6, 10, 15, 18, 22, 29 and 45 after the initiation of treatment
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 5 | 9
hours | NA [0.8 to NA] — No median estimate was obtained due to the small group sizes and the small number of events assessed. | 6.0 [0.3 to NA] — No CI estimate was obtained due to the small group sizes and the small number of events assessed. | NA [1.5 to NA] — No median estimate was obtained due to the small group sizes and the small number of events assessed. | NA [0.8 to NA] — No median estimate was obtained due to the small group sizes and the small number of events assessed. | 8.0 [4.0 to NA] — No CI estimate was obtained due to the small group sizes and the small number of events assessed. | 47.3 [0.8 to NA] — No CI estimate was obtained due to the small group sizes and the small number of events assessed.
Statistical Analysis 1: Comparison: RPH - 20 mg vs Voltaren® (Diclofenac); Test type: Other; p = 0.5995, Log Rank
Statistical Analysis 2: Comparison: RPH - 160 mg vs Voltaren® (Diclofenac); Test type: Other; p = 0.9012, Log Rank

9. Secondary Outcome: Time to Use of the Rescue Medication
Description: Time to use of the rescue medication was calculated as the time in hours from the date/time of administration (first dose) of the investigational product to the date/time of the first use of the rescue medication.
Time Frame: from the date/time of IP administration (first dose) to the date/time of the first use of the rescue medication, up to day 60
Population: Patient 01003 was excluded from the analysis of the endpoint due to the use of prohibited therapy (methylprednisolone 125 mg, IV, daily from the 2nd day of therapy until the end of the study).
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac)
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 5 | 9
hours | 23.7 [21.3 to 24.5] | NA [3.1 to NA] — No median estimate was obtained due to the small group sizes and the small number of events assessed. | 71.8 [24.4 to NA] — No CI estimate was obtained due to the small group sizes and the small number of events assessed. | 84.6 [22.7 to NA] — No CI estimate was obtained due to the small group sizes and the small number of events assessed. | NA [3.0 to NA] — No median estimate was obtained due to the small group sizes and the small number of events assessed. | NA [4.4 to NA] — No median estimate was obtained due to the small group sizes and the small number of events assessed.

10. Secondary Outcome: Proportion of Patients Who Received a Rescue Therapy Agent
Description: The proportion of patients who received the rescue medication within 72 hours of starting the investigational product therapy
Time Frame: 72 hours after the initiation of treatment with the test drug
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac)
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 5 | 9
Participants | 12 | 1 | 3 | 3 | 2 | 2
Statistical Analysis 1: Comparison: RPH - 4 mg vs Voltaren® (Diclofenac); Test type: Other; p = 0.0066, Fisher Exact; difference in proportions = 63.5, 95% CI 2-sided [19.9 to 88.6]
Statistical Analysis 2: Comparison: RPH - 20 mg vs Voltaren® (Diclofenac); Test type: Other; p > 0.9999, Fisher Exact; difference in proportions = -5.6, 95% CI 2-sided [-50.1 to 45.5]
Statistical Analysis 3: Comparison: RPH - 40 mg vs Voltaren® (Diclofenac); Test type: Other; p = 0.3287, Fisher Exact; difference in proportions = 27.8, 95% CI 2-sided [-26.8 to 71.8]
Statistical Analysis 4: Comparison: RPH - 80 mg vs Voltaren® (Diclofenac); Test type: Other; p = 0.3287, Fisher Exact; difference in proportions = 27.8, 95% CI 2-sided [-26.8 to 71.8]
Statistical Analysis 5: Comparison: RPH - 160 mg vs Voltaren® (Diclofenac); Test type: Other; p = 0.5804, Fisher Exact; difference in proportions = 17.8, 95% CI 2-sided [-33.7 to 67.8]

11. Secondary Outcome: Proportion of Patients Who Received a Rescue Therapy Agent
Description: The proportion of patients who received the rescue medication over the entire treatment period
Time Frame: up to day 60
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac)
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 5 | 9
Participants | 13 | 1 | 4 | 4 | 2 | 3

12. Secondary Outcome: Changes in the Health Assessment Questionnaire (HAQ) Parameters: Disability Index
Description: Changes in the Health Assessment Questionnaire (HAQ) parameters in 15, 29 and 45 days following the initiation of treatment with the test drug as compared to baseline.
  (The result for each of the 8 categories ("Dressing and Grooming", "Arising", "Eating", "Walking", "Hygiene", "Reach", "Grip", "Activities") of the HAQ questionnaire was calculated as the maximum score of responses (on an ordinal scale from 0 (best) to 3 (worst): without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3)) to questions included in this category. If the patient required outside help or any of the specified aids or devices to perform actions related to a certain category, then this category was assigned "2" points, if the point was not equal to "3", i.e. points "0" and "1" increased to "2". The sum of points for the evaluated categories was calculated and divided by the number of categories, which gives a disability index in the range of 0 to 3.)
Time Frame: Baseline and 15, 29 and 45 days following the initiation of treatment with the test drug
Population: It should be noted that estimates following the use of the rescue medication or a prohibited analgesic were not included in the descriptive statistics.
Measure: Mean (Standard Deviation); unit: units of the HAQ index
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 5 | 9
units of the HAQ index
  Baseline value | 1.3 (0.802) | 1.23 (0.578) | 1.75 (0.806) | 1.1 (0.649) | 1.6 (0.615) | 1.32 (0.577)
  Change Day 15: number analyzed (Participants) | 1 | 4 | 1 | 1 | 2 | 6
  Change Day 15 | -0.75 (NA) — small group size | -0.63 (0.685) | -0.88 (NA) — small group size | -0.63 (NA) — small group size | -1.06 (0.619) | -0.56 (0.342)
  Change Day 29: number analyzed (Participants) | 1 | 4 | 1 | 1 | 2 | 4
  Change Day 29 | -0.13 (NA) — small group size | -1.09 (0.672) | -1.25 (NA) — small group size | -0.63 (NA) — small group size | -0.5 (0.53) | -0.38 (0.144)
  Change Day 45: number analyzed (Participants) | 1 | 3 | 1 | 1 | 2 | 4
  Change Day 45 | -0.38 (NA) — small group size | -1.42 (0.382) | -1.38 (NA) — small group size | -0.63 (NA) — small group size | -0.56 (0.619) | -0.44 (0.298)

13. Other Pre Specified Outcome: Pharmacokinetics (PK) - Area Under the Plasma concentration-of RPH-104 Under the Subcutaneous Administration
Description: Including area under the plasma concentration-time curve over the dosing interval (AUC0-tau)
Time Frame: Baseline and in 2,8,24,48,72 hours,on Days 5,6,10,15,18,22,29,45 following the initiation of treatment with the test drug and on the follow-up visit (in case of premature withdrawal of patient)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg
Number analyzed (Participants) | 15 | 5 | 6 | 5 | 3
h*ng/mL | 38000 (124) | 762000 (152) | 845000 (45) | 1620000 (36.5) | 3230000 (38.2)

14. Other Pre Specified Outcome: Pharmacokinetics (PK) - Area Under the Active Substance Concentration- of RPH-104 Under the Subcutaneous Administration
Description: Including Area under the active substance concentration-time curve from zero (before drug administration) to infinity (AUC0-∞)
Time Frame: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg
Number analyzed (Participants) | 14 | 5 | 6 | 5 | 3
h*ng/mL | 47900 (97.9) | 816000 (155) | 901000 (44.3) | 1720000 (37.1) | 3380000 (38.1)

15. Other Pre Specified Outcome: Pharmacokinetics (PK) - Maximum Concentration of the Active Substance -of RPH-104 Under the Subcutaneous Administration
Description: Including Maximum concentration of the active substance (Cmax)
Time Frame: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg
Number analyzed (Participants) | 15 | 5 | 6 | 6 | 4
ng/mL | 142 (110) | 2220 (155) | 2380 (47.7) | 4860 (18) | 9760 (38.2)

16. Other Pre Specified Outcome: Pharmacokinetics (PK) of RPH-104 Under the Subcutaneous Administration
Description: Including elimination constant (Kel)
Time Frame: as for outcome 13
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg
Number analyzed (Participants) | 14 | 5 | 6 | 5 | 3
1/h | 0.00298 (0.000573) | 0.00314 (0.000622) | 0.00304 (0.000241) | 0.00317 (0.000575) | 0.00294 (0.000311)

17. Other Pre Specified Outcome: Pharmacokinetics (PK) -Time to Reach Maximum Concentration of the Active Substance - of RPH-104 Under the Subcutaneous Administration
Description: Including Time to reach maximum concentration of the active substance (tmax)
Time Frame: as for outcome 13
Measure: Median (Full Range); unit: hours
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg
Number analyzed (Participants) | 15 | 5 | 6 | 6 | 4
hours | 93.7 [8 to 120] | 47.5 [21.3 to 72.1] | 84.8 [47.1 to 120] | 82.7 [24 to 122] | 94.4 [72 to 96.1]

18. Other Pre Specified Outcome: Pharmacokinetics (PK) - Terminal Half-life -of RPH-104 Under the Subcutaneous Administration
Description: Including terminal half-life (T 1/2)
Time Frame: as for outcome 13
Measure: Median (Full Range); unit: hours
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg
Number analyzed (Participants) | 14 | 5 | 6 | 5 | 3
hours | 248 [153 to 285] | 235 [170 to 274] | 223 [205 to 256] | 231 [168 to 264] | 241 [212 to 261]

19. Other Pre Specified Outcome: Change in the Serum Rate of High-sensitive CRP (Hs-CRP) in Specified Timeframes
Description: Change in the serum rate of high-sensitive CRP (hs-CRP) in 24, 72 hours, on Days 5, 6, 15, 29 and 45 following the initiation of treatment with the test drug compared to baseline
Time Frame: Baseline and in 24, 72 hours, on Days 5, 6, 15, 29 and 45 after the initiation of treatment with the test drug
Population: Number of valid observations is presented.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 5 | 9
mg/L
  Baseline value | 36.673 (31.3545) | 8.295 (6.6212) | 10.105 (14.2834) | 37.908 (25.5594) | 35.396 (32.4800) | 15.769 (18.0878)
  Day 2/ 24 hours: number analyzed (Participants) | 14 | 5 | 6 | 5 | 4 | 9
  Day 2/ 24 hours | 35.468 (32.2025) | 20.338 (33.3728) | 24.483 (16.3543) | 28.864 (16.1194) | 12.000 (11.5518) | 22.716 (26.9958)
  Day 4/ 72 hours: number analyzed (Participants) | 15 | 5 | 6 | 5 | 4 | 9
  Day 4/ 72 hours | 33.894 (35.0873) | 3.408 (0.8120) | 12.900 (9.3579) | 11.846 (6.1780) | 8.678 (10.5037) | 9.279 (8.1642)
  Day 5: number analyzed (Participants) | 15 | 4 | 6 | 5 | 4 | 9
  Day 5 | 32.279 (32.6858) | 3.090 (0.9076) | 7.142 (5.7071) | 8.696 (3.6468) | 6.178 (6.4262) | 8.877 (6.3308)
  Day 6: number analyzed (Participants) | 15 | 4 | 6 | 5 | 4 | 9
  Day 6 | 29.065 (28.1288) | 2.710 (1.6140) | 3.650 (2.8445) | 4.604 (1.3871) | 3.190 (3.0165) | 8.417 (7.0440)
  Day 15: number analyzed (Participants) | 13 | 5 | 5 | 4 | 5 | 9
  Day 15 | 21.017 (28.4384) | 2.642 (1.4322) | 3.304 (5.8018) | 5.115 (3.5382) | 4.042 (6.1199) | 6.579 (4.4134)
  Day 29: number analyzed (Participants) | 15 | 5 | 6 | 5 | 4 | 8
  Day 29 | 16.811 (26.3922) | 7.532 (13.0615) | 2.750 (2.9068) | 5.014 (2.8480) | 10.998 (17.3463) | 7.595 (7.9870)
  Day 45 | 24.958 (29.4450) | 3.570 (2.1907) | 2.445 (1.8315) | 3.093 (0.5652) | 14.500 (19.2882) | 11.734 (11.4627)

20. Other Pre Specified Outcome: Change in the Rate of Serum Amyloid Protein A in the Specified Timeframes
Description: Change in the rate of serum amyloid protein A in 24, 72 hours and on Day 5, 6, 15, 29 and 45 following the initiation of treatment with the test drug as compared to baseline
Time Frame: Baseline and in 24, 72 hours and on Day 5, 6, 15, 29 and 45 following the initiation of treatment with the test drug
Population: Number of valid observations is presented.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 5 | 9
ng/mL
  Baseline value: number analyzed (Participants) | 13 | 5 | 6 | 4 | 4 | 8
  Baseline value | 13493.687 (14565.0449) | 2516.606 (1367.7981) | 16764.020 (14525.1072) | 16168.130 (12937.7377) | 16291.605 (17949.6741) | 5033.151 (3384.3761)
  Day 2/ 24 hours: number analyzed (Participants) | 15 | 4 | 6 | 5 | 4 | 9
  Day 2/ 24 hours | 17424.060 (17167.2073) | 11078.300 (19281.3822) | 20104.555 (15608.3760) | 15581.486 (13271.7115) | 3659.778 (3244.2099) | 7294.631 (5163.5001)
  Day 4/ 72 hours: number analyzed (Participants) | 15 | 4 | 6 | 4 | 4 | 9
  Day 4/ 72 hours | 17588.735 (16623.4301) | 1171.203 (400.3851) | 12162.612 (12060.2753) | 14419.760 (11828.2546) | 10596.423 (16813.3253) | 7362.322 (9834.7459)
  Day 5: number analyzed (Participants) | 15 | 4 | 6 | 5 | 4 | 9
  Day 5 | 17360.201 (15874.5237) | 1195.975 (393.6981) | 5680.190 (5708.9022) | 8228.272 (7624.1329) | 5952.460 (10455.6856) | 8252.633 (8121.6203)
  Day 6: number analyzed (Participants) | 15 | 4 | 6 | 5 | 3 | 9
  Day 6 | 18553.955 (15454.2373) | 1847.923 (1646.0125) | 4781.173 (6120.5728) | 5799.608 (5562.9980) | 6117.777 (8569.9756) | 6165.779 (5356.4841)
  Day 15: number analyzed (Participants) | 13 | 5 | 5 | 4 | 4 | 8
  Day 15 | 9272.782 (11297.9676) | 1525.612 (502.8845) | 8899.982 (17399.0042) | 4582.338 (5995.5993) | 2732.598 (1325.3698) | 6031.146 (10261.9489)
  Day 29: number analyzed (Participants) | 15 | 5 | 6 | 5 | 3 | 8
  Day 29 | 8918.439 (12001.1492) | 4255.756 (6845.1947) | 1645.107 (1044.8811) | 3626.702 (2740.1283) | 3618.843 (3147.2319) | 3779.410 (2727.9500)
  Day 45: number analyzed (Participants) | 15 | 4 | 6 | 3 | 3 | 7
  Day 45 | 13858.845 (16512.5575) | 2086.198 (2799.5039) | 1269.680 (695.3511) | 1567.040 (1421.4541) | 9885.230 (15228.9607) | 7289.553 (7189.8429)

21. Other Pre Specified Outcome: Change in the Serum Rates of Cytokines: IL-1α
Description: Change in the serum rates of IL-1α in 24, 72 hours and on Days 5, 6, 15, 29 and 45 following the initiation of treatment with the test drug as compared to baseline
Time Frame: Baseline and in 24, 72 hours and on Days 5, 6, 15, 29 and 45 following the initiation of treatment with the test drug
Population: Number of valid observations is presented. (IL-1a values <1.10 were replaced with 1.09 for graphical representation and statistical analysis.)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 5 | 9
pg/mL
  Baseline value: number analyzed (Participants) | 13 | 6 | 6 | 6 | 5 | 9
  Baseline value | 1.090 (0.0000) | 1.090 (0.0000) | 1.090 (0.0000) | 1.752 (1.5390) | 1.090 (0.0000) | 1.090 (0.0000)
  Day 2/ 24 hours: number analyzed (Participants) | 15 | 5 | 6 | 5 | 4 | 9
  Day 2/ 24 hours | 1.090 (0.0000) | 1.090 (0.0000) | 1.097 (0.0163) | 1.782 (1.5474) | 1.090 (0.0000) | 1.090 (0.0000)
  Day 4/ 72 hours: number analyzed (Participants) | 15 | 5 | 6 | 5 | 4 | 9
  Day 4/ 72 hours | 1.090 (0.0000) | 1.090 (0.0000) | 1.090 (0.0000) | 1.688 (1.3372) | 1.090 (0.0000) | 1.090 (0.0000)
  Day 5: number analyzed (Participants) | 15 | 4 | 6 | 5 | 4 | 9
  Day 5 | 1.090 (0.0000) | 1.090 (0.0000) | 1.090 (0.0000) | 1.790 (1.5652) | 1.090 (0.0000) | 1.090 (0.0000)
  Day 6: number analyzed (Participants) | 15 | 4 | 6 | 5 | 4 | 9
  Day 6 | 1.090 (0.0000) | 1.090 (0.0000) | 1.090 (0.0000) | 1.612 (1.1672) | 1.090 (0.0000) | 1.090 (0.0000)
  Day 15: number analyzed (Participants) | 13 | 5 | 5 | 4 | 5 | 9
  Day 15 | 1.132 (0.1525) | 1.090 (0.0000) | 1.090 (0.0000) | 1.090 (0.0000) | 1.090 (0.0000) | 1.090 (0.0000)
  Day 29: number analyzed (Participants) | 15 | 5 | 6 | 5 | 4 | 8
  Day 29 | 1.097 (0.0258) | 1.090 (0.0000) | 1.090 (0.0000) | 1.090 (0.0000) | 1.090 (0.0000) | 1.090 (0.0000)
  Day 45: number analyzed (Participants) | 15 | 4 | 6 | 3 | 3 | 7
  Day 45 | 1.090 (0.0000) | 1.090 (0.0000) | 1.090 (0.0000) | 1.090 (0.0000) | 1.090 (0.0000) | 1.090 (0.0000)

22. Other Pre Specified Outcome: Change in the Serum Rates of Cytokines: IL-1β
Description: Change in the serum rates of IL-1β in 24, 72 hours and on Days 5, 6, 15, 29 and 45 following the initiation of treatment with the test drug as compared to baseline
Time Frame: Baseline and in 24, 72 hours and on Days 5, 6, 15, 29 and 45 following the initiation of treatment with the test drug
Population: Number of valid observations is presented. (IL-1β <0.30 values were replaced with 0.29, IL-1β > 500.00 values were replaced with 500.01 for graphical presentation and statistical analysis.)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 5 | 9
pg/mL
  Baseline value: number analyzed (Participants) | 13 | 6 | 6 | 6 | 5 | 9
  Baseline value | 39.035 (138.5078) | 1.080 (1.9351) | 0.290 (0.0000) | 2.558 (3.5248) | 0.290 (0.0000) | 0.290 (0.0000)
  Day 2/ 24 hours: number analyzed (Participants) | 15 | 5 | 6 | 5 | 4 | 9
  Day 2/ 24 hours | 33.885 (128.9519) | 0.290 (0.0000) | 0.290 (0.0000) | 1.100 (1.8112) | 0.290 (0.0000) | 0.290 (0.0000)
  Day 4/ 72 hours: number analyzed (Participants) | 15 | 5 | 6 | 5 | 4 | 9
  Day 4/ 72 hours | 33.759 (128.9859) | 0.290 (0.0000) | 0.290 (0.0000) | 2.112 (4.0741) | 0.290 (0.0000) | 0.290 (0.0000)
  Day 5: number analyzed (Participants) | 15 | 4 | 6 | 5 | 4 | 9
  Day 5 | 33.753 (128.9873) | 0.290 (0.0000) | 0.290 (0.0000) | 0.290 (0.0000) | 0.290 (0.0000) | 0.290 (0.0000)
  Day 6: number analyzed (Participants) | 15 | 4 | 6 | 5 | 4 | 9
  Day 6 | 33.998 (128.9231) | 0.290 (0.0000) | 0.290 (0.0000) | 2.362 (4.6331) | 0.290 (0.0000) | 0.290 (0.0000)
  Day 15: number analyzed (Participants) | 13 | 5 | 5 | 4 | 5 | 9
  Day 15 | 38.730 (138.5974) | 1.222 (2.0840) | 0.290 (0.0000) | 1.965 (3.3500) | 0.290 (0.0000) | 0.290 (0.0000)
  Day 29: number analyzed (Participants) | 15 | 5 | 6 | 5 | 4 | 8
  Day 29 | 33.811 (128.9724) | 1.320 (2.3032) | 0.417 (0.3103) | 1.746 (3.2557) | 0.290 (0.0000) | 0.290 (0.0000)
  Day 45: number analyzed (Participants) | 15 | 4 | 6 | 3 | 3 | 7
  Day 45 | 0.290 (0.0000) | 0.290 (0.0000) | 0.290 (0.0000) | 0.290 (0.0000) | 0.290 (0.0000) | 0.290 (0.0000)

23. Other Pre Specified Outcome: Change in the Serum Rates of Cytokines: Interleukin -1 Receptor Antagonist (IL-1RA)
Description: Change in the serum rates of IL-1RA in 24, 72 hours and on Days 5, 6, 15, 29 and 45 following the initiation of treatment with the test drug as compared to baseline
Time Frame: Baseline and in 24, 72 hours and on Days 5, 6, 15, 29 and 45 following the initiation of treatment with the test drug
Population: Number of valid observations is presented. (IL-1RA values <30.00 were replaced with 29.99 for graphical representation and statistical analysis.)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 5 | 9
pg/mL
  Baseline value: number analyzed (Participants) | 13 | 6 | 6 | 6 | 5 | 9
  Baseline value | 2400.500 (1495.1100) | 1448.978 (527.8658) | 1671.010 (1225.2673) | 2240.155 (937.1988) | 2619.456 (2706.3397) | 2090.721 (1240.5717)
  Day 2/ 24 hours: number analyzed (Participants) | 15 | 5 | 6 | 5 | 4 | 9
  Day 2/ 24 hours | 1700.180 (1448.4981) | 229.842 (291.9887) | 153.098 (145.3780) | 29.990 (0.0000) | 29.990 (0.0000) | 2483.891 (1786.0361)
  Day 4/ 72 hours: number analyzed (Participants) | 15 | 5 | 6 | 5 | 4 | 9
  Day 4/ 72 hours | 1295.743 (916.8659) | 156.216 (110.6281) | 140.108 (123.8956) | 157.654 (227.2334) | 29.990 (0.0000) | 2297.651 (1361.7429)
  Day 5: number analyzed (Participants) | 15 | 4 | 6 | 5 | 4 | 9
  Day 5 | 1364.993 (1106.8245) | 187.223 (109.9846) | 154.463 (124.6690) | 87.214 (79.7269) | 29.990 (0.0000) | 2417.991 (1416.8428)
  Day 6: number analyzed (Participants) | 15 | 4 | 6 | 5 | 4 | 9
  Day 6 | 1407.230 (927.8243) | 214.610 (125.9518) | 203.688 (133.0562) | 180.492 (112.2664) | 29.990 (0.0000) | 2426.761 (1452.6687)
  Day 15: number analyzed (Participants) | 13 | 5 | 5 | 4 | 5 | 9
  Day 15 | 1620.332 (935.4363) | 374.900 (96.9459) | 474.542 (214.5880) | 645.085 (300.6542) | 257.492 (166.0738) | 2249.794 (1459.3243)
  Day 29: number analyzed (Participants) | 15 | 5 | 6 | 5 | 4 | 8
  Day 29 | 1928.417 (1048.0875) | 563.892 (142.6097) | 583.062 (269.1237) | 686.992 (305.9470) | 471.178 (267.8262) | 1870.815 (1032.8765)
  Day 45: number analyzed (Participants) | 15 | 4 | 6 | 3 | 3 | 7
  Day 45 | 1806.647 (858.8185) | 915.010 (177.2813) | 808.212 (354.6509) | 711.997 (285.9941) | 518.063 (201.1455) | 1969.547 (1352.6193)

24. Other Pre Specified Outcome: Change in the Serum Rates of Cytokines: IL-6
Description: Change in the serum rates of IL-6 in 24, 72 hours and on Days 5, 6, 15, 29 and 45 following the initiation of treatment with the test drug as compared to baseline
Time Frame: Baseline and in 24, 72 hours and on Days 5, 6, 15, 29 and 45 following the initiation of treatment with the test drug
Population: Number of valid observations is presented. (IL-6 values <0.92 were replaced with 0.913, IL-6 values >200.00 were replaced with 200.01 for graphical representation and statistical analysis.)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 5 | 9
pg/mL
  Baseline value: number analyzed (Participants) | 13 | 6 | 6 | 6 | 5 | 9
  Baseline value | 26.035 (39.1257) | 5.005 (4.6022) | 34.307 (54.3264) | 5.623 (6.8564) | 13.666 (11.9695) | 6.058 (6.9686)
  Day 2/ 24 hours: number analyzed (Participants) | 15 | 5 | 6 | 5 | 4 | 9
  Day 2/ 24 hours | 27.030 (42.9908) | 2.084 (1.8930) | 37.788 (72.3187) | 6.284 (11.1153) | 9.065 (12.5843) | 2.361 (1.2039)
  Day 4/ 72 hours: number analyzed (Participants) | 15 | 5 | 6 | 5 | 4 | 9
  Day 4/ 72 hours | 14.943 (29.9008) | 2.236 (1.8533) | 2.145 (0.9961) | 3.142 (3.7290) | 4.698 (7.3223) | 1.702 (1.1067)
  Day 5: number analyzed (Participants) | 15 | 4 | 6 | 5 | 4 | 9
  Day 5 | 23.999 (37.5678) | 2.695 (2.2949) | 2.378 (1.9432) | 1.396 (0.5031) | 4.905 (7.5114) | 1.823 (1.6473)
  Day 6: number analyzed (Participants) | 15 | 4 | 6 | 5 | 4 | 9
  Day 6 | 8.391 (13.3742) | 3.565 (3.5282) | 2.965 (3.4991) | 1.272 (0.3636) | 6.220 (9.8491) | 2.157 (2.1250)
  Day 15: number analyzed (Participants) | 13 | 5 | 5 | 4 | 5 | 9
  Day 15 | 10.595 (14.4444) | 2.870 (1.5838) | 2.434 (1.7929) | 1.793 (0.5907) | 12.858 (25.3149) | 2.036 (1.2089)
  Day 29: number analyzed (Participants) | 15 | 5 | 6 | 5 | 4 | 8
  Day 29 | 18.643 (50.4658) | 2.758 (1.7315) | 3.278 (4.2245) | 1.482 (0.5334) | 17.903 (31.1335) | 5.304 (7.4387)
  Day 45: number analyzed (Participants) | 15 | 4 | 6 | 3 | 3 | 7
  Day 45 | 6.466 (9.1261) | 4.608 (5.8999) | 3.370 (4.5051) | 1.537 (0.3911) | 3.753 (1.6094) | 2.607 (1.9663)

25. Other Pre Specified Outcome: Change in the Serum Rates of Cytokines: IL-8
Description: Change in the serum rates of IL-8 in 24, 72 hours and on Days 5, 6, 15, 29 and 45 following the initiation of treatment with the test drug as compared to baseline
Time Frame: Baseline and in 24, 72 hours and on Days 5, 6, 15, 29 and 45 following the initiation of treatment with the test drug
Population: Number of valid observations is presented. (IL-8 values <2.00 were replaced with 1.99 for graphical representation and statistical analysis.)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 5 | 9
pg/mL
  Baseline value: number analyzed (Participants) | 13 | 5 | 6 | 6 | 5 | 8
  Baseline value | 12.384 (5.8297) | 21.964 (24.8759) | 9.277 (4.5347) | 18.305 (21.8921) | 12.318 (12.5702) | 10.863 (7.1505)
  Day 2/ 24 hours: number analyzed (Participants) | 15 | 5 | 6 | 5 | 4 | 9
  Day 2/ 24 hours | 8.228 (7.1217) | 9.304 (9.7609) | 9.030 (5.5014) | 12.304 (9.9136) | 2.668 (1.3550) | 17.141 (13.6494)
  Day 4/ 72 hours: number analyzed (Participants) | 15 | 4 | 6 | 5 | 4 | 9
  Day 4/ 72 hours | 15.601 (19.4714) | 8.708 (5.8951) | 9.020 (6.2030) | 5.952 (4.4991) | 8.148 (5.6025) | 15.980 (11.7350)
  Day 5: number analyzed (Participants) | 15 | 4 | 6 | 5 | 4 | 9
  Day 5 | 13.521 (7.8988) | 4.313 (2.6941) | 8.032 (4.9402) | 10.518 (6.8098) | 11.190 (4.4376) | 15.188 (12.3696)
  Day 6: number analyzed (Participants) | 15 | 4 | 6 | 5 | 4 | 9
  Day 6 | 16.969 (16.9723) | 8.015 (4.6897) | 7.937 (5.3199) | 7.594 (5.9449) | 10.745 (6.3010) | 19.881 (21.0673)
  Day 15: number analyzed (Participants) | 13 | 5 | 5 | 4 | 5 | 9
  Day 15 | 9.765 (9.3536) | 20.884 (31.6507) | 11.520 (7.4313) | 16.395 (19.5556) | 3.060 (2.3926) | 34.770 (66.4033)
  Day 29: number analyzed (Participants) | 15 | 5 | 6 | 5 | 4 | 8
  Day 29 | 19.766 (20.8879) | 25.622 (36.4743) | 8.003 (6.1368) | 8.596 (9.2114) | 9.243 (5.1441) | 8.554 (7.6207)
  Day 45: number analyzed (Participants) | 15 | 4 | 6 | 3 | 3 | 7
  Day 45 | 12.664 (7.2467) | 5.468 (4.1120) | 5.807 (5.8272) | 7.223 (3.0891) | 7.927 (5.3051) | 11.763 (11.1239)

26. Other Pre Specified Outcome: Change in the Serum Rates of Cytokines: Tumor Necrosis Factor (TNF-α)
Description: Change in the serum rates of TNF-α in 24, 72 hours and on Days 5, 6, 15, 29 and 45 following the initiation of treatment with the test drug as compared to baseline
Time Frame: Baseline and in 24, 72 hours and on Days 5, 6, 15, 29 and 45 following the initiation of treatment with the test drug
Population: Number of valid observations is presented. (TNF-α values <2.30 were replaced with 2.29 for graphical representation and statistical analysis.)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 5 | 9
pg/mL
  Baseline value: number analyzed (Participants) | 13 | 6 | 6 | 6 | 5 | 9
  Baseline value | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000)
  Day 2/ 24 hours: number analyzed (Participants) | 15 | 5 | 6 | 5 | 4 | 9
  Day 2/ 24 hours | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000)
  Day 4/ 72 hours: number analyzed (Participants) | 15 | 4 | 6 | 5 | 4 | 9
  Day 4/ 72 hours | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000)
  Day 5: number analyzed (Participants) | 15 | 4 | 6 | 5 | 4 | 9
  Day 5 | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000)
  Day 6: number analyzed (Participants) | 15 | 4 | 6 | 5 | 4 | 9
  Day 6 | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000)
  Day 15: number analyzed (Participants) | 13 | 5 | 5 | 4 | 5 | 9
  Day 15 | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000)
  Day 29: number analyzed (Participants) | 15 | 5 | 6 | 5 | 4 | 8
  Day 29 | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000)
  Day 45: number analyzed (Participants) | 15 | 4 | 6 | 3 | 3 | 7
  Day 45 | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000) | 2.290 (0.0000)

27. Secondary Outcome: Changes in the Health Assessment Questionnaire (HAQ) Parameters: Arising
Description: Changes in the Health Assessment Questionnaire (HAQ) parameters in 15, 29 and 45 days following the initiation of treatment with the test drug as compared to baseline.
  The result was calculated as the maximum score of responses (on an ordinal scale from 0 to 3) to questions included in this category. Patients were asked about their ability to complete these tasks in the past week using the following categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 (best) to 3 (worst).
  If the patient required outside help or any of the specified aids or devices to perform actions related to a certain category, then this category was assigned "2" points, if the point was not equal to "3", i.e. points "0" and "1" increased to "2".
Time Frame: Baseline and 15, 29 and 45 days following the initiation of treatment with the test drug
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units of the HAQ index
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 5 | 9
units of the HAQ index
  Baseline value | 0.9 (0.74) | 1.3 (0.52) | 1.5 (1.05) | 0.7 (0.82) | 1.4 (0.55) | 1.2 (0.97)
  Change Day 15: number analyzed (Participants) | 1 | 4 | 1 | 1 | 2 | 6
  Change Day 15 | -1.0 (NA) — small group size | -1.0 (0.82) | -1.0 (NA) — small group size | 0.0 (NA) — small group size | -1.0 (0.00) | -0.5 (0.55)
  Change Day 29: number analyzed (Participants) | 1 | 4 | 1 | 1 | 2 | 4
  Change Day 29 | -1.0 (NA) — small group size | -1.3 (0.50) | -1.0 (NA) — small group size | 0.0 (NA) — small group size | -0.5 (0.71) | 0.0 (0.82)
  Change Day 45: number analyzed (Participants) | 1 | 3 | 1 | 1 | 2 | 4
  Change Day 45 | -1.0 (NA) — small group size | -1.3 (0.58) | -1.0 (NA) — small group size | 0.0 (NA) — small group size | -0.5 (0.71) | 0.0 (0.0)

28. Secondary Outcome: Changes in the Health Assessment Questionnaire (HAQ) Parameters: Eating
Description: as for outcome 27
Time Frame: Baseline and 15, 29 and 45 days following the initiation of treatment with the test drug
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units of the HAQ index
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 5 | 9
units of the HAQ index
  Baseline value | 1.0 (1.20) | 0.7 (0.82) | 1.3 (1.37) | 0.8 (1.17) | 1.0 (1.00) | 0.7 (1.00)
  Change Day 15: number analyzed (Participants) | 1 | 4 | 1 | 1 | 2 | 6
  Change Day 15 | 0.0 (NA) — small group size | -0.5 (1.0) | 0.0 (NA) — small group size | 0.0 (NA) — small group size | 0.0 (0.00) | -0.3 (0.52)
  Change Day 29: number analyzed (Participants) | 1 | 4 | 1 | 1 | 2 | 4
  Change Day 29 | 0.0 (NA) — small group size | -1.0 (0.82) | 0.0 (NA) — small group size | 0.0 (NA) — small group size | -0.5 (0.71) | -0.3 (0.50)
  Change Day 45: number analyzed (Participants) | 1 | 3 | 1 | 1 | 2 | 4
  Change Day 45 | 0.0 (NA) — small group size | -1.3 (0.58) | 0.0 (NA) — small group size | 0.0 (NA) — small group size | -0.5 (0.71) | -0.3 (0.5)

29. Secondary Outcome: Changes in the Health Assessment Questionnaire (HAQ) Parameters: Walking
Description: as for outcome 27
Time Frame: Baseline and 15, 29 and 45 days following the initiation of treatment with the test drug
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units of the HAQ index
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 5 | 9
units of the HAQ index
  Baseline value | 1.4 (0.74) | 1.8 (0.75) | 1.8 (1.17) | 1.3 (0.82) | 1.6 (1.14) | 1.8 (0.67)
  Change Day 15: number analyzed (Participants) | 1 | 4 | 1 | 1 | 2 | 6
  Change Day 15 | 0.0 (NA) — small group size | -1.3 (0.96) | -1.0 (NA) — small group size | -1.0 (NA) — small group size | -1.5 (0.71) | -0.7 (0.82)
  Change Day 29: number analyzed (Participants) | 1 | 4 | 1 | 1 | 2 | 4
  Change Day 29 | 0.0 (NA) — small group size | -1.3 (0.96) | -2.0 (NA) — small group size | -1.0 (NA) — small group size | -0.5 (0.71) | -0.3 (0.50)
  Change Day 45: number analyzed (Participants) | 1 | 3 | 1 | 1 | 2 | 4
  Change Day 45 | 0.0 (NA) — small group size | -1.3 (1.15) | -2.0 (NA) — small group size | -1.0 (NA) — small group size | -0.5 (0.71) | -0.8 (0.96)

30. Secondary Outcome: Changes in the Health Assessment Questionnaire (HAQ) Parameters: Hygiene
Description: as for outcome 27
Time Frame: Baseline and 15, 29 and 45 days following the initiation of treatment with the test drug
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units of the HAQ index
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 5 | 9
units of the HAQ index
  Baseline value | 1.2 (1.21) | 1.2 (0.98) | 1.7 (1.03) | 1.5 (1.05) | 2.2 (0.45) | 1.3 (0.50)
  Change Day 15: number analyzed (Participants) | 1 | 4 | 1 | 1 | 2 | 6
  Change Day 15 | -1.0 (NA) — small group size | -0.3 (1.26) | -1.0 (NA) — small group size | -1.0 (NA) — small group size | -2.5 (0.71) | -0.5 (0.55)
  Change Day 29: number analyzed (Participants) | 1 | 4 | 1 | 1 | 2 | 4
  Change Day 29 | 1.0 (NA) — small group size | -1.3 (0.96) | -1.0 (NA) — small group size | -1.0 (NA) — small group size | -0.5 (0.71) | -0.5 (0.58)
  Change Day 45: number analyzed (Participants) | 1 | 3 | 1 | 1 | 2 | 4
  Change Day 45 | 0.0 (NA) — small group size | -1.7 (0.58) | -1.0 (NA) — small group size | -1.0 (NA) — small group size | -0.5 (0.71) | -1.0 (0.82)

31. Secondary Outcome: Changes in the Health Assessment Questionnaire (HAQ) Parameters: Grip
Description: as for outcome 27
Time Frame: Baseline and 15, 29 and 45 days following the initiation of treatment with the test drug
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units of the HAQ index
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac)
Number analyzed (Participants) | 15 | 6 | 6 | 6 | 5 | 9
units of the HAQ index
  Baseline value | 1.4 (0.99) | 1.0 (0.63) | 1.2 (1.17) | 1.0 (1.10) | 1.2 (1.10) | 0.4 (0.73)
  Change Day 15: number analyzed (Participants) | 1 | 4 | 1 | 1 | 2 | 6
  Change Day 15 | -1.0 (NA) — small group size | -0.5 (0.58) | 0.0 (NA) — small group size | -1.0 (NA) — small group size | 0.0 (0.00) | -0.2 (0.41)
  Change Day 29: number analyzed (Participants) | 1 | 4 | 1 | 1 | 2 | 4
  Change Day 29 | -1.0 (NA) — small group size | -1.0 (0.82) | 0.0 (NA) — small group size | -1.0 (NA) — small group size | -0.5 (0.71) | -0.3 (0.5)
  Change Day 45: number analyzed (Participants) | 1 | 3 | 1 | 1 | 2 | 4
  Change Day 45 | -1.0 (NA) — small group size | -1.3 (0.58) | 0.0 (NA) — small group size | -1.0 (NA) — small group size | -1.0 (1.41) | 0.3 (1.26)

ADVERSE EVENTS:
Time Frame: The safety of the investigational product was assessed over a 60-day period of therapy and follow-up. The tables show AEs that developed from the start of therapy.
Description: The safety population included all subjects who received at least one dose of the investigational product. This population was used for all treatment safety assessments. The safety analysis of data was performed based on the actual treatment received by the patients.
Arm/Group | RPH - 4 mg | RPH - 20 mg | RPH - 40 mg | RPH - 80 mg | RPH - 160 mg | Voltaren® (Diclofenac)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/6 | 0/6 | 0/6 | 0/5 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/6 | 0/6 | 2/6 | 0/5 | 1/9
Other Adverse Events (participants affected / at risk) | 11/15 | 1/6 | 3/6 | 3/6 | 4/5 | 2/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RPH - 4 mg (N=15) | RPH - 20 mg (N=6) | RPH - 40 mg (N=6) | RPH - 80 mg (N=6) | RPH - 160 mg (N=5) | Voltaren® (Diclofenac) (N=9)
drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mycobacterium tuberculosis complex test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RPH - 4 mg (N=15) | RPH - 20 mg (N=6) | RPH - 40 mg (N=6) | RPH - 80 mg (N=6) | RPH - 160 mg (N=5) | Voltaren® (Diclofenac) (N=9)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal scarring (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Administration site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Genitourinary chlamydia infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mycoplasma infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureaplasma infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mycobacterium tuberculosis complex test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil percentage decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Joint swelling (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Daydreaming (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Micturition disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study related information could be made public available only after Sponsors written permission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/92/NCT04067492/Prot_SAP_000.pdf